CLINICAL TRIAL: NCT06560125
Title: Clinical Study to Evaluate the Performance of WOUNDCHEK Bacterial Status With Trained vs Untrained Users
Brief Title: WOUNDCHEK Bacterial Status Performance With Trained vs Untrained Users
Status: Completed | Type: Observational
Sponsor: Woundchek Laboratories BV (Industry)
Responsible Party: Sponsor
Other Study IDs: PROT-2023-001/004
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2024-08

CONDITIONS: Wound
MeSH Terms: conditions — Wounds and Injuries | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- WOUNDCHEK Bacterial Status positive: Wounds testing positive for bacterial protease activity
  Interventions: Other: Standard care
- WOUNDCHEK Bacterial Status negative: Wounds testing negative for bacterial protease activity
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Standard care — Treatment appropriate for wound condition

SUMMARY:
The purpose of this clinical study is to evaluate the performance of WOUNDCHEK™ Bacterial Status (WCBS) with untrained users in diverse CLIA waived locations and trained users and compare the results to those obtained in the study used for De Novo approval (DEN180014). Untrained and trained users are as defined in the FDA guidance document entitled 'Recommendations for Clinical Laboratory Improvement Amendments of 1988 (CLIA) Waiver Applications for Manufacturers of In Vitro Diagnostic Devices' (Feb 2020). The test result will be blinded to the clinician treating the wound. The healing outcome at 12 weeks following the test will be compared for wounds positive vs negative for bacterial protease activity (BPA). Study success criteria will be that the positive likelihood ratio (PLR) of a BPA positive wound being non-healing at 12 weeks for both trained and untrained users will be statistically comparable to the PLR obtained in the study submitted for DEN180014.

DETAILED DESCRIPTION:
WCBS is an in vitro diagnostic chromatographic test for the qualitative detection of bacterial protease activity directly from wound fluid samples collected with a swab. The WCBS test is intended for use in adult patients as an aid in assessing the risk for non-healing of chronic venous, diabetic foot, and pressure ulcers associated with wounds where there are no signs of wound infection and where patients are asymptomatic for clinical signs of infection. The test is intended for use with chronic wounds that are between 21 days and < 6 months of age and chronic wounds that are ≥ 6 months of age that are < 1cm2 in size. This test is indicated for use solely by health care professionals whose clinical practice primarily or routinely involves the assessment and treatment of chronic wounds. WCBS results are intended for use in conjunction with the assessment of other known risk factors for wound healing that significantly contribute to the risk for non-healing chronic wounds such as wound age, wound size, and vascular status.

This is a prospective study designed to evaluate the performance of WCBS by testing wound fluid swab samples collected from leg ulcers (LU), diabetic foot ulcers (DFU), and pressure ulcers (PU) in waived environments that represent the device's intended user locations by untrained users compared to trained users in environments certified to perform CLIA moderate complexity tests.

At the time of a Subject's initial study enrolment (Day 0), one wound fluid swab sample will be collected from the designated wound area of each Subject from whom informed consent has been obtained. All swab specimens will be collected using swabs provided with the test kit. For the purpose of this study, this swab will be tested at the time of collection on the WCBS test by clinical site staff members, according to product instructions.

All WCBS test operators will not be the treating clinician. Throughout the study, all health care providers responsible for treatment of the Subjects, will be blinded to the WCBS test results.

Over the course of the 12 weeks post Day 0, Subjects will be treated per each site's Standard of Care. For the purposes of this study, clinical healing status, determined by whether or not the wound has achieved complete closure over a 12-week time frame will be utilized as the primary "comparator method" for evaluation of device performance. A WCBS negative test result on a wound determined to be "healed" at or before the "Week 12" time point will be considered a "true negative". A WCBS positive test result on a wound determined to be "not healed" by the "Week 12" time point will be considered a "true positive". For wounds not healed by 12 weeks, the percent wound area reduction over the 12 week period will be calculated.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has presented to the participating study site with a VLU, DFU and / or a PU that is suspected not to be infected, as determined by the Investigator and/ or study staff - defined as one that does not show more than two of the NERDS signs of infection.
2. Subject is 18 years of age or older.
3. The wound is between 21 days and 6 months of age or more than 6 months of age if less than 1cm2 in area.
4. Subject agrees to complete all aspects of the study and provides written Informed Consent per IRB requirements.

Exclusion Criteria:

1. Subject does not meet inclusion criteria.
2. The wound is less than 21 days of age or more than six months if larger than 1cm2 in area.
3. Topical antimicrobial treatment will be started on the target wound at the time of subject enrollment. Note: Specific treatment used will be left to the PI's discretion.
4. Topical antimicrobial treatment is being used on the target wound at the time of subject enrollment, and the treatment will be continued. Note: Specific treatment used will be left to the PI's discretion.
5. Target wound contains a malignancy.
6. Subject has hypersensitivity of the wound or painful wound surface which prevents touching/swabbing of the wound surface.
7. Subject is confirmed to be positive for HIV or hepatitis.
8. Subject is unable or unwilling to provide informed consent.
9. A designated wound area may only be enrolled once in the study. For example, if an enrolled wound heals to complete closure and then re-opens, it cannot be re-enrolled in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects attending wound clinic
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-12-24 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Wound healing | 12 weeks
  Complete wound closure

SECONDARY OUTCOMES:
Wound size reduction | 12 weeks
  Percent change in wound size

CONTACTS AND LOCATIONS:
Overall Officials: Aliza Lee, DPM, Principal Investigator — Salem VA
Locations (1):
- Salem VA Medical Centre, Salem, Virginia, United States